CLINICAL TRIAL: NCT06275386
Title: Drug-Coated Balloon in Native Chronic Total Occlusion Percutaneous Coronary Intervention (IMAGINATION)
Brief Title: Drug-Coated Balloon in Native Chronic Total Occlusion Percutaneous Coronary Intervention
Acronym: IMAGINATION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.31/II/24
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease; Total Occlusion of Coronary Artery
Keywords: chronic total occlusion; percutaneous coronary intervention; drug-coated balloon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug-coated balloon (Experimental): Patients will undergo PCI of the native coronary CTO with a DCB.
  Interventions: Device: Paclitaxel Drug-coated balloon

INTERVENTIONS:
Device: Paclitaxel Drug-coated balloon — Percutaneous coronary intervention of the actual CTO body with a paclitaxel drug-coated balloon.

SUMMARY:
The IMAGINATION trial is an investigator-initiated, prospective, single-center study of symptomatic patients with a native chronic total occlusion (CTO) undergoing intravascular ultrasound (IVUS)-guided percutaneous coronary intervention (PCI) with a drug-coated balloon (DCB). Post-PCI IVUS and fractional flow reserve (FFR) at baseline and at 6-months follow-up will be performed. In addition, patients included in the coronary computed tomography angiography (CCTA) substudy will undergo CCTA at 12-months follow-up. The aim of this study is to evaluate the efficacy and safety of DCB-only approach in native coronary CTO.

DETAILED DESCRIPTION:
Whereas CTO PCI techniques and success rates have significantly improved during the last decade, CTOs still pose a significant technical challenge for accurate stent sizing (primarily due to negative remodelling and subsequent distal vessel dilatation post-PCI) resulting in a potentially increased risk of stent failure. Hence, the concept of DCB as a definitive treatment for native CTO is appealing and warrants further investigation. The IMAGINATION trial has been designed as a prospective research to: 1) investigate both the immediate and intermediate-term angiographic, IVUS and physiologic efficacy outcomes as well as safety profile of DCB for native vessel coronary CTO, and 2) to provide a basis for future randomized clinical trial comparing DCB to drug-eluting stents.

All patients with CTO will be screened for potential inclusion in the study. After obtaining written informed consent, patients with successful intraplaque guidewire crossing through CTO lesion (excluding the use of dissection and re-entry techniques) will undergo IVUS-guided PCI with a scoring balloon (balloon-to-artery ratio of 1:1) followed by the use of a paclitaxel-coated balloon. Following satisfactory angiographic result, IVUS and physiological measurements (FFR and non-hyperemic pressure ratios) in the target vessel will be performed. At 6-months follow-up, invasive angiography with IVUS and FFR/non-hyperemic pressure ratios in the target vessel will be repeated. In addition, patients with pre-procedural CCTA will undergo follow-up CCTA after 12 months (CCTA substudy).

ELIGIBILITY:
Inclusion Criteria:

* clinical indication for CTO PCI as determined by the local heart team (presence of angina or equivalent symptoms and/or documented ischemia or viability)
* native CTO lesion as defined by invasive coronary angiography
* informed consent for participation in the study

Exclusion Criteria:

* <18 years of age
* myocardial infarction
* cardiogenic shock
* severe valvular disease
* estimated life expectancy <1 year
* contraindication to PCI
* positive pregnancy test or breast-feeding
* in-stent CTO
* CTO recanalization using antegrade or retrograde dissection and re-entry techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
In-segment late lumen loss | 6-months
  The difference by subtracting the minimal lumen diameter (MLD) at follow-up from the MLD postprocedure. In-segment equals DCB plus the proximal and distal 5-mm margins.

SECONDARY OUTCOMES:
Angiographic outcomes assessed directly post-PCI | immediately post-procedure (1 day)
  * minimum lumen diameter (mm)
  * residual diameter stenosis (%)
  * the rate of bail-out stenting after DCB use (%)
HD-IVUS outcomes assessed directly post-PCI | immediately post-procedure (1 day)
  * minimal lumen diameter (mm)
  * minimal lumen area (mm2)
  * maximum plaque burden (%)
Physiologic outcomes assessed directly post-PCI | immediately post-procedure (1 day)
  * the ratio of pd/pa
  * cRR (absolute values)
  * FFR (absolute values)
Angiographic outcomes at 6-months follow-up | 6-months
  * minimum lumen diameter (mm)
  * residual diameter stenosis (%)
  * in-segment binary restenosis (≥50% diameter stenosis)
  * the rate of target vessel re-occlusion (yes/no)
HD-IVUS outcomes at 6-months follow-up | 6-months
  * minimal lumen diameter (mm)
  * minimal lumen area (mm2)
  * maximum plaque burden (%)
Physiologic outcomes at 6-months follow-up | 6-months
  * the ratio of pd/pa
  * cRR (absolute values)
  * FFR (absolute values)
Computed tomographic outcomes at 12-months follow-up (CCTA substudy) | 12-months
  * minimal lumen area (mm2)
  * maximum plaque burden (%)
  * area stenosis (%)
  * diameter stenosis (%)
  * remodeling index (absolute values)
  * total plaque volume (mm3)
  * calcified plaque volume (mm3)
  * non-calcified plaque volume (mm3)
  * low-attenuation plaque volume (mm3)
  * percentage of change in in-segment total plaque volume (%)
  * percentage of change in in-segment calcified plaque volume (%)
  * percentage of change in in-segment non-calcified plaque volume (%)
  * percentage of change in in-segment low-attenuation plaque volume (%)
  * percentage of change in in-segment remodeling index (%)
Clinical outcomes at 12-months follow-up | 12-months
  • the rate of target lesion failure (composite endpoint of cardiac death, target vessel-related myocardial infarction, or clinically-driven target lesion revascularization)

CONTACTS AND LOCATIONS:
Overall Officials: Maksymilian Opolski, Principal Investigator — National Institute of Cardiology
Locations (1):
- National Institute of Cardiology, Warsaw, Masovian Voivodeship, Poland